CLINICAL TRIAL: NCT02775942
Title: Safety and Immunogenicity of an Inactivated Poliomyelitis Vaccine (IPOVAC) in Vietnamese Children
Brief Title: Safety and Immunogenicity of IPOVAC in Young Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Ministry of Science and Technology, Vietnam (Other Government)
Responsible Party: Principal Investigator, Dang Duc Anh, General Director, National Institute of Hygiene and Epidemiology, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-IPOVAC-02
Record Dates: First submitted 2016-05-05; First posted 2016-05-18 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2016-05

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IPOVAC 1.5:5:5 (Experimental): IPOVAC- POLYVAC Vietnam Composition: Type 1: 1.5DU, Type 2: 5DU, Type 3:5DU Subcutaneous inj 0.5ml/dose, 3 doses, interval 30days +/- 3 days Liquid form
  Interventions: Biological: IPOVAC 1.5:5:5
- IPOVAC 3:10:10 (Experimental): IPOVAC- POLYVAC Vietnam Composition: Type 1: 3DU, Type 2: 10DU, Type 3:10DU Subcutaneous inj 0.5ml/dose, 3 doses, interval 30days +/- 3 days Liquid form
  Interventions: Biological: IPOVAC, 3:10:10
- IPOVAC 6:20:20 (Experimental): IPOVAC- POLYVAC Vietnam Composition: Type 1: 6DU, Type 2: 20DU, Type 3:20DU Subcutaneous inj 0.5ml/dose, 3 doses, interval 30days +/- 3 days Liquid form
  Interventions: Biological: IPOVAC, 6:20:20
- IMOVAC-POLIO (Active Comparator): IMOVAC-POLIO (Sanofi Pasteur), liquid form composition: Type 1 (Mahoney) 40DU, Type 2 (MEF1) 8DU, Type 3 (Saukett) 32 DU, Subcutaneous route 0.5ml/dose, 3 doses, 4-week interval
  Interventions: Biological: IMOVAC-POLIO

INTERVENTIONS:
Biological: IMOVAC-POLIO — IMOVAC-POLIO (Sanofi Pasteur), liquid form composition: Type 1 (Mahoney) 40DU, Type 2 (MEF1) 8DU, Type 3 (Saukett) 32 DU, Subcutaneous route 0.5ml/dose, 3 doses, 4-week interval
  Other Names: IMOVAC
  Arms: IMOVAC-POLIO
Biological: IPOVAC 1.5:5:5 — IPOVAC- POLYVAC Vietnam Composition: Type 1: 1.5DU, Type 2: 5DU, Type 3:5DU Subcutaneous inj 0.5ml/dose, 3 doses, interval 30days +/- 3 days Liquid form
  Other Names: IPOVAC-low
  Arms: IPOVAC 1.5:5:5
Biological: IPOVAC, 3:10:10 — IPOVAC- POLYVAC Vietnam Composition: Type 1: 3DU, Type 2: 10DU, Type 3:10DU Subcutaneous inj 0.5ml/dose, 3 doses, interval 30days +/- 3 days Liquid form
  Other Names: IPOVAC-medium
  Arms: IPOVAC 3:10:10
Biological: IPOVAC, 6:20:20 — IPOVAC- POLYVAC Vietnam Composition: Type 1: 6DU, Type 2: 20DU, Type 3:20DU Subcutaneous inj 0.5ml/dose, 3 doses, interval 30days +/- 3 days Liquid form
  Other Names: IPOVAC-high
  Arms: IPOVAC 6:20:20

SUMMARY:
A dose escalating study with 3 different dosing regimens of the studied vaccine (IPOVAC- POLYVAC-Vietnam) and a licensed vaccine (IMOVAC-Sanofi Pasteur- France) is conducted in Vietnamese children, aged 2 months and above to assess the safety and immunogenicity. Two hundred and forty children are enrolled and placed randomly into 4 groups (60 children/group), each of which receive 3 doses of vaccine subcutaneously, at 4 week interval. Safety issues included immediate reaction at the site of injection and systemic reaction within 30 min of administration, within 7 days after each dose, unexpected event occur within 30 days of each dose, SAE (from start of dose 1 to 30 days after dose 3), blood cell count, urea, ALT,AST. Immunogenicity outcomes include seroconversion of neutralising antibodies for each of vaccine serotypes.

DETAILED DESCRIPTION:
The use of oral poliomyelitis vaccine (OPV) in Vietnam expanded immunisation program has resulted in successful eradication of polio in Vietnam. However due to the concern of OPV-related poliomyelitis cases occurred worldwide, WHO has recommended the countries to gradually change to inactivated polio vaccine (IPV). In Vietnam, POLYVAC has been approved and sponsored by the Ministry of Science and Technology to produce IPV under Japanese technology. The vaccine consisting of 3 serotypes (Serotype 1,2 and 3) has been proven safety in volunteer adults.

In this study, a dose escalating study with 3 different dosing regimens of the studied vaccine (IPOVAC) and a licensed vaccine (IMOVAC-Sanofi Pasteur- France) is conducted in Vietnamese children, aged 2 months and above to assess the safety and immunogenicity. Two hundred and forty children are enrolled and placed randomly into 4 groups (60 children/group), each of which receive 3 doses of vaccine subcutaneously, at 4 week interval. Safety issues evaluated include immediate reaction at the site of injection and systemic reaction within 30 min of administration, within 7 days after each dose, unexpected event occur within 30 days of each dose, SAE (from start of dose 1 to 30 days after dose 3), blood cell count, urea, ALT,AST. Seroconversion rates of neutralising antibodies for each of vaccine serotypes are to be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, 2 months of ages
* Full term babies (>=37 weeks)
* Weight at birth (>=2500gr)
* Have not been vaccinated with polio vaccine or vaccine containing poliovirus components
* Not currently have acute infection (assessed via clinical check up and asking parents/care givers about health history before enrolment
* Parents/legal guardians agree to participate their children in this study and sign the informed consent.

Exclusion Criteria:

* Currently have chronic diseases (cardiovascular, liver and spleen related etc)
* Use (orally or through infection) with corticoid containing drug (>1mg/kg dose)
* Use of immunocompromised treatment within 4 weeks of enrolment
* Being immunocompromised and autoimmune diseases (HIV, lupus)
* the history of immunocompromised in the family
* history of high fever
* Allergic for any vaccine component
* Fever (>38oC) within 3 days before vaccination or at enrolment
* Malnourished (3rd level or above)
* Blood disorder
* use of vaccines which have not been licences 7 days before enrolment in this study

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07-25 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events after each dose of vaccine | Upto 30 days after each dose
  Number of participants with treatment-related adverse events after each dose of vaccine, immediately after vaccination (within 30 min), within 7 days and 30 days of vaccination, as assessed by CTCAE v.4.0
Number of participants with 4-fold or more increase in in antibody titers after 2 or 3 doses of vaccine (compared to pre-vaccination) | Upto 30 days after the final dose
  Seroconversion rate of each IPOVAC regimen and IMOVAC after 2 or 3 doses of vaccines

SECONDARY OUTCOMES:
Number of participants with treatment-related SAE after each vaccination dose | Upto 30 days after vaccine dose
  Number of participants with treatment-related SAE after each vaccination doses of IPOVAC compared to that of IMOVAC, as assessed by CTCAE ver 4.0
Number of participants with abnormal laboratory value | Upto 30 days after each vaccine dose
  Numbers of participants with abnormal laboratory values (blood cell counts, urea concentration, liver function (ALT, AST concentration) when administered with different IPOVAC formulations and with IMOVAC before and after each dose of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Dang D Anh, PhD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (2):
- Vietnam (2):
  - Preventive Medicine center, Thanh Sơn, Phu Tho
  - Phu Tho Preventive Medicine Center, Việt Trì, Phu Tho

IPD SHARING:
Plan to Share IPD: No
Individual data with identification removed are to be available for Ethical committee, Ministry of Health and National Foundation of Science and Technology Development to avoid misuse of data.
  Public shared data will be in the form of summarised tables and figures.